CLINICAL TRIAL: NCT02627833
Title: Lungfunction, Lung Clearance Index, Bronchial Inflammation and Epigenetics of Patients With Bronchiolitis Obliterans
Brief Title: Lung Function, LCI, Bronchial Inflammation and Epigenetics of Patients With BO
Acronym: FRABO-03
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Rosewich, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: MRosewich
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Bronchiolitis Obliterans
Keywords: induced Sputum; lung clearance index; miRNA; inflammation; chronic lung disease
MeSH Terms: conditions — Bronchiolitis Obliterans; Inflammation | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cells of induced Sputum, blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subject Group: Patients suffering from Bronchiolitis Obliterans
  Interventions: Other: observation
- Control Group: Age and sex matched control group
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — Record lung function, Lung clearance index, inflammatory status

SUMMARY:
Bronchiolitis obliterans is a chronic disease in which a persistent inflammatory process leads to obliteration of the small airways. Pulmonary function tests (body plethysmography with DLCO, lung clearance index) are performed and the fraction of exhaled nitric oxide is measured. A blood test is following to determine the inflammatory status und collect miRNA. Induced Sputum will be obtained.

DETAILED DESCRIPTION:
The purpose of this study is to compare miRNA pattern, lung function values, bronchial inflammation and the Lung clearance index of Patients with Bronchiolitis obliterans aged between 6 up to 30 years of age with a matched control group.

The sputum samples will be processed and quantitatively analyzed to get a profile of the cytological composition.

Sputum and serum samples are analyzed by quantitative real-time polymerase chain reaction (qRT-PCR) and by cytometric bead assay (CBA). miRNA samples will be collected, processand compared with the miRNA database at http://www.mirbase.org/

Methods and Work Programme:

* Measurement of nitric oxide in expired air (FeNO)
* Lung function testing with spirometry and body plethysmography
* Lung clearance index (LCI)
* Bronchodilation
* Blood test: blood count, CRP, RAST, serum inflammatory mediators, (genetic markers of the non-specific pulmonary defense system), miRNA analysis
* Induced sputum for inflammatory mediators and microbiological investigations

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age between 6 an 35 years
* known bronchiolitis obliterans (Group Bronchiolitis)/ no Bronchiolitis Obliterans (Group matched controls)
* ability to perform lung function tests and inhale correctly

Exclusion Criteria:

* <6 years of age
* >35 years of age
* acute systemic or bronchial inflammation
* other chronic diseases or infection (e.g. HIV, Tbc, malignoma)
* pregnancy
* alcohol, drug or illegal drug abuse
* disability to register the range and consequences of the study
* actual participation in another study

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with the assured diagnose of Bronchiolitis Obliterans and controls without this disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
miRNA Status | single day observation
  Blood sample to determine candidate miRNA for Bronchiolitis obliterans

OTHER OUTCOMES:
Lung clearance index (LCI) | single day observation
  Determine Lung clearance index with the Oxygen washout method
FVC [%-pred.] | single day observation
  Compare FVC [%-pred.] of BO Patients with a healthy control group
FEV1 [%-pred.] | single day observation
  Compare FEV1[%-pred.] of BO Patients with a healthy control group
Tiffeneau Index | single day observation
  Compare Tiffeneau-Index of BO Patients with a healthy control group
sRtot [%-pred.] | single day observation
  Compare sRtot[%-pred.] of BO Patients with a healthy control group
RV/TLC [%-pred.] | single day observation
  Compare RV/TLC[%-pred.] of BO Patients with a healthy control group
DLCO [%-pred.] | single day observation
  Compare difffusion capacity of the lung for CO [%-pred.] of BO Patients with a healthy control group
IL-6 (pg/ml) | single day observation
  Comparing IL-6 in Serum of patients with BO with a healthy control group
IL-8 (pg/ml | single day observation
  Comparing IL-8 in Serum of patients with BO with a healthy control group
Il-17 (pg/ml) | single day observation
  Comparing IL-17 in Serum of patients with BO with a healthy control group
CrP (mg/dl) | single day observation
  Comparing CrP in Serum of patients with BO with a healthy control group
FeNO ppb | single day observation
  Comparing FeNO in exhaled air of patients with BO with a healthy control group
Sputum cell count | single day observation
  Comparing sputum cell counts of patients with BO with a healthy control group

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rosewich, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Kurland G, Michelson P. Bronchiolitis obliterans in children. Pediatr Pulmonol. 2005 Mar;39(3):193-208. doi: 10.1002/ppul.20145. PMID 15635614
- [Background] Boehler A, Kesten S, Weder W, Speich R. Bronchiolitis obliterans after lung transplantation: a review. Chest. 1998 Nov;114(5):1411-26. doi: 10.1378/chest.114.5.1411. No abstract available. PMID 9824023
- [Background] Moonnumakal SP, Fan LL. Bronchiolitis obliterans in children. Curr Opin Pediatr. 2008 Jun;20(3):272-8. doi: 10.1097/MOP.0b013e3282ff62e9. PMID 18475095
- [Result] Pichler M, Herrmann G, Schmidt H, Ahrens P, Zielen S. Persistent adenoviral infection and chronic obstructive bronchitis in children: is there a link? Pediatr Pulmonol. 2001 Nov;32(5):367-71. doi: 10.1002/ppul.1145. PMID 11596161
- [Result] Rosewich M, Zissler UM, Kheiri T, Voss S, Eickmeier O, Schulze J, Herrmann E, Ducker RP, Schubert R, Zielen S. Airway inflammation in children and adolescents with bronchiolitis obliterans. Cytokine. 2015 May;73(1):156-62. doi: 10.1016/j.cyto.2014.10.026. Epub 2015 Mar 6. PMID 25748838
- [Result] Motameny S, Wolters S, Nurnberg P, Schumacher B. Next Generation Sequencing of miRNAs - Strategies, Resources and Methods. Genes (Basel). 2010 Jun 3;1(1):70-84. doi: 10.3390/genes1010070. PMID 24710011